CLINICAL TRIAL: NCT00286182
Title: Efficacy of Treating Anemia in Heart Failure With a Preserved Ejection Fraction (HFPEF) on Ventricular Function, Exercise Capacity and Health Status
Brief Title: Anemia in Heart Failure With a Preserved Ejection Fraction (HFPEF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mathew S. Maurer (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Mathew S. Maurer, Associate Professor of Clinical Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAB3037; R01AG027518-01 (NIH)
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Anemia
Keywords: Heart Failure; Elderly; Diastolic Dysfunction; Anemia; Ventricular End Diastolic Volume; Aged
MeSH Terms: conditions — Anemia; Heart Failure | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin alpha (Experimental): Subcutaneous erythropoietin will be administered once weekly to achieve a target hemoglobin of 13 g/dL. Subjects will be dosed with the study drug for 24 weeks. The administration of study drug will be performed according to a pre-specified treatment algorithm that adjust erythropoietin dosages based on the rate of rise of the hemoglobin.
  Interventions: Drug: Erythropoietin alpha
- Placebo (Placebo Comparator): Placebo consists of saline injections.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erythropoietin alpha — Erythropoietin alpha is administered weekly by subcutaneous injection using a pre-specified dosing algorithm. The dosing algorithm is designed to make adjustments based on the rate of rise (ROR) of the hemoglobin over a one week period, as well as the absolute hemoglobin value. Subjects initially received active treatment with 7,500 units of erythropoietin given weekly by subcutaneously injection. Subjects are carefully monitored (e.g. every week) to avoid rapid increases in hemoglobin/hematocrit and/or increasing blood pressure control. Dose adjustments are made if the hemoglobin rises too rapidly (greater than 0.3 g/dL) in any given weekly interval.
  Other Names: Erythropoietin alpha (Epogen)
  Arms: Erythropoietin alpha
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if treating anemia with subcutaneous erythropoetin in patients with heart failure and a preserved ejection fraction (HFPEF) will be associated with reverse ventricular remodeling, significant improvements in exercise capacity, and improved health status, as compared with placebo.

DETAILED DESCRIPTION:
Heart failure frequently occurs in patients with a preserved ejection fraction (HFPEF) and affected subjects are predominantly elderly women with several co-morbid conditions. Despite the diversity of underlying clinical pathologies and co-morbid conditions present in these patients, a common pathophysiologic explanation is generally applied to explain their clinical symptoms. Our preliminary data show that a significant subgroup with HFPEF has increases in ventricular volumes and expanded plasma volumes, consistent with a volume overloaded state. In the setting of a preserved EF with end diastolic volume increased, stroke volume must increase, indicating a high output state. Anemia may be an important, modifiable contributor to the observed high output and volume overload as well as exercise intolerance in elderly HFPEF patients, abnormal ventricular remodeling and impaired overall health status and quality of life. This protocol evaluates the impact of treating anemia in subjects with HFPEF. The specific aims of the current study are to provide a comprehensive and mechanistically based assessment of how correcting anemia in subjects with HFPEF can impact on functional capacity, ventricular structure and function and overall health status. We propose to perform a randomized, prospective, double blind study in 80 subjects with HFPEF to test the hypothesis that the administration of subcutaneous erythropoietin will be associated with reverse ventricular remodeling, significant improvements in exercise capacity and improved health status.

ELIGIBILITY:
Inclusion Criteria:

1. Heart failure and a preserved ejection fraction (HFPEF) - EF >=40%
2. Anemia - defined as hemoglobin < 12 g/dL
3. Age >= 55 years
4. Patients must be able to understand and sign the informed consent document after the nature of the study has been fully explained, prior to beginning any study procedures.

Exclusion Criteria:

1. Presence of uncontrolled hypertension (Systolic blood pressure > 160 mm Hg and/or diastolic blood pressure > 90 mm Hg)
2. Resting heart rate > 120 bpm
3. Baseline 6-minute walk test > 450 meters
4. Valvular heart disease (e.g. more than mild regurgitant or stenotic mitral, aortic, tricuspid, or pulmonic valve disease).
5. Infiltrative cardiac disease such as hemochromatosis and amyloidosis
6. Hypertrophic cardiomyopathy
7. Chronic pulmonary disease (FEV 1 < 60% predicted)
8. Renal failure (GFR < 15 ml/min)
9. Hemoglobin < 8 g/dL
10. BMI > 40
11. Exercise limited by angina, claudication, orthopedic, or neurological diseases.
12. Severe liver dysfunction that is defined by an international normalized ratio > 2.0, not caused by an anticoagulant.
13. Current or recent treatment (within past 6 months) with erythropoietin
14. Erythropoietin level > 100 mU/ml
15. Recent cardiac surgery (< 3 months)
16. Known iron deficiency anemia from chronic GI blood loss, uterine bleeding, or other chronic bleeding
17. Planned surgery during the course of the study
18. Significant alcohol use or illicit drug use.
19. Patients with a known hypercoagulable state.
20. Active hematologic disease (e.g. sickle cell anemia, thalassemia, chronic myelogenous leukemia) or malignancy
21. Patients with current seizure disorder or activity
22. Patients who are known to be pregnant
23. History of deep venous thrombosis (DVT) or pulmonary embolus (PE) within 12 months before study entry. Prior superficial thrombophlebitis is not an exclusion criterion.
24. History of cerebrovascular accident (CVA) within 6 months
25. History of transient ischemic attack (TIA) within 6 months
26. History of acute coronary syndrome (ACS), or other arterial thrombosis within 6 months before study entry. ACS includes unstable angina, Q wave myocardial infarction (QwMI), and non-Q wave myocardial infarction (NQMI).
27. Allergy or sensitivity to human serum albumin
28. Known hypersensitivity to mammalian cell-derived products

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew S Maurer, MD, Principal Investigator — Columbia University
Locations (1):
- Clinical Cardiovascular Research Laboratory for the Elderly, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maurer MS, King DL, El-Khoury Rumbarger L, Packer M, Burkhoff D. Left heart failure with a normal ejection fraction: identification of different pathophysiologic mechanisms. J Card Fail. 2005 Apr;11(3):177-87. doi: 10.1016/j.cardfail.2004.10.006. PMID 15812744
- [Background] Brucks S, Little WC, Chao T, Rideman RL, Upadhya B, Wesley-Farrington D, Sane DC. Relation of anemia to diastolic heart failure and the effect on outcome. Am J Cardiol. 2004 Apr 15;93(8):1055-7. doi: 10.1016/j.amjcard.2003.12.062. PMID 15081458
- [Background] Silverberg DS, Wexler D, Blum M, Tchebiner J, Sheps D, Keren G, Schwartz D, Baruch R, Yachnin T, Shaked M, Zubkov A, Steinbruch S, Iaina A. The correction of anemia in severe resistant heart failure with erythropoietin and intravenous iron prevents the progression of both the heart and the renal failure and markedly reduces hospitalization. Clin Nephrol. 2002 Jul;58 Suppl 1:S37-45. PMID 12227725
- [Background] Silverberg DS, Wexler D, Sheps D, Blum M, Keren G, Baruch R, Schwartz D, Yachnin T, Steinbruch S, Shapira I, Laniado S, Iaina A. The effect of correction of mild anemia in severe, resistant congestive heart failure using subcutaneous erythropoietin and intravenous iron: a randomized controlled study. J Am Coll Cardiol. 2001 Jun 1;37(7):1775-80. doi: 10.1016/s0735-1097(01)01248-7. PMID 11401110
- [Background] Mancini DM, Katz SD, Lang CC, LaManca J, Hudaihed A, Androne AS. Effect of erythropoietin on exercise capacity in patients with moderate to severe chronic heart failure. Circulation. 2003 Jan 21;107(2):294-9. doi: 10.1161/01.cir.0000044914.42696.6a. PMID 12538431
- [Background] Klapholz M, Maurer M, Lowe AM, Messineo F, Meisner JS, Mitchell J, Kalman J, Phillips RA, Steingart R, Brown EJ Jr, Berkowitz R, Moskowitz R, Soni A, Mancini D, Bijou R, Sehhat K, Varshneya N, Kukin M, Katz SD, Sleeper LA, Le Jemtel TH; New York Heart Failure Consortium. Hospitalization for heart failure in the presence of a normal left ventricular ejection fraction: results of the New York Heart Failure Registry. J Am Coll Cardiol. 2004 Apr 21;43(8):1432-8. doi: 10.1016/j.jacc.2003.11.040. PMID 15093880
- [Derived] Green P, Babu BA, Teruya S, Helmke S, Prince M, Maurer MS. Impact of epoetin alfa on left ventricular structure, function, and pressure volume relations as assessed by cardiac magnetic resonance: the heart failure preserved ejection fraction (HFPEF) anemia trial. Congest Heart Fail. 2013 Jul-Aug;19(4):172-9. doi: 10.1111/chf.12027. Epub 2013 Mar 20. PMID 23517485
- [Derived] Maurer MS, Teruya S, Chakraborty B, Helmke S, Mancini D. Treating anemia in older adults with heart failure with a preserved ejection fraction with epoetin alfa: single-blind randomized clinical trial of safety and efficacy. Circ Heart Fail. 2013 Mar;6(2):254-63. doi: 10.1161/CIRCHEARTFAILURE.112.969717. Epub 2012 Dec 20. PMID 23258574
- [Derived] Altincatal A, Macarthur RB, Teruya S, Helmke S, Maurer MS. A dosing algorithm for erythropoietin alpha in older adults with heart failure and a preserved ejection fraction. Cardiovasc Ther. 2013 Apr;31(2):92-9. doi: 10.1111/j.1755-5922.2011.00295.x. Epub 2011 Aug 26. PMID 21884028

RESULTS

PARTICIPANT FLOW:
Groups:
- Erythropoietin Alpha: Subcutaneous erythropoietin will be administered once weekly to achieve a target hemoglobin of 13 g/dL. Subjects will be dosed with the study drug for 24 weeks. The administration of study drug will be performed according to a pre-specified treatment algorithm that adjust erythropoietin dosages based on the rate of rise of the hemoglobin.
  Erythropoietin alpha: Erythropoietin alpha is administered weekly by subcutaneous injection using a pre-specified dosing algorithm. The dosing algorithm is designed to make adjustments based on the rate of rise (ROR) of the hemoglobin over a one week period, as well as the absolute hemoglobin value. Subjects initially received active treatment with 7,500 units of erythropoietin given weekly by subcutaneously injection. Subjects are carefully monitored (e.g. every week) to avoid rapid increases in hemoglobin/hematocrit and/or increasing blood pressure control. Dose adjustments are made if the hemoglobin rises too rapidly (greater than 0.3 g/dL) in
Period: Overall Study
Arm/Group | Erythropoietin Alpha | Placebo
Started | 28 | 28
Completed | 23 | 25
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erythropoietin Alpha | Placebo | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 79 (11) | 74 (9) | 76.5 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular End-diastolic Volume
Description: This outcome measure is collected using a three dimensional echocardiography.
Time Frame: Baseline and 6 month
Measure: Mean (Standard Error); unit: mL
Arm/Group | Erythropoietin Alpha | Placebo
Number analyzed (Participants) | 23 | 25
mL | -6 (14) | -4 (16)

ADVERSE EVENTS:
Arm/Group | Erythropoietin Alpha | Placebo
Serious Adverse Events (participants affected / at risk) | 19/28 | 18/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erythropoietin Alpha (N=28) | Placebo (N=28)
Hospitalization (General disorders) | 16 (16) | 14 (14)
Sudden Death (General disorders) | 0 (0) | 1 (1) — Sudden death unrelated to the treatment: Subject was vacationing and collapsed on a beach and died suddenly. No cause of death was determined.
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 3 (3) | 2 (2) — Hospitalized

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes